CLINICAL TRIAL: NCT06135103
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Hybrid Decentralized Study to Evaluate the Safety and Efficacy of Daily Subcutaneous (SC) Injection of TXA127 in Post-ischemic Stroke Patients
Brief Title: Phase 2 Study of TXA127 in Post-ischemic Stroke Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Constant Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXA127-STRK-001
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- talfirastide (TXA127) (Experimental): TXA127 will be given daily for 12 weeks at a dose of 0.5.mg/kg via SC injection.
  Interventions: Drug: talfirastide
- placebo (Placebo Comparator): Placebo will be given daily for 12 weeks via SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: talfirastide — TXA127, a pharmaceutically formulated angiotensin (1-7) heptapeptide, identical to the endogenously produced, non-hypertensive derivative of angiotensin II (Ang II) is a sterile solution containing angiotensin (1-7) [A(1-7)], supplied in a 3 mL, single-use, stoppered vial.
  Other Names: TXA127
  Arms: talfirastide (TXA127)
Drug: Placebo — Placebo is a sterile solution containing supplied in a 3 mL, single-use, stoppered vial.
  Arms: placebo

SUMMARY:
This is a 50-patient, Phase 2, double-blind, randomized, placebo-controlled, hybrid decentralized study to evaluate the safety and efficacy of daily subcutaneous (SC) injection of TXA127 in post-ischemic stroke patients. Subjects will receive either TXA127 0.5mg/kg or placebo for 12 weeks started 6 to 24 months post ischemic stroke, and they will have a 12 week follow up visit after treatment has ended. The primary efficacy outcome measure is individual patient absolute change from baseline in motor and sensory functions as measured by the Fugl-Meyer Assessment of Upper Extremity (FMA-UE) 12 weeks after start of treatment.

DETAILED DESCRIPTION:
This is a safety, tolerability, and efficacy study in patients with sensorimotor deficits after confirmed middle cerebral artery ischemic stroke. The study will be double-blinded and placebo-controlled and conducted over a period of approximately 6 months, with treatment starting 6-24 months after stroke. After obtaining informed consent, eligibility will be determined by review of medical history and assessments of patient's condition. To establish a baseline, all assessments will be completed prior to administration of the first dose of study drug.

Patients will be randomized (1:1) to receive either subcutaneous (SC) placebo or TXA127 (0.5 mg/kg) injections once daily for 12 weeks. In addition to receiving either the study drug or placebo, patients will be required to undergo physical therapy (PT) or occupational therapy (OT) at least twice a week. Patients will be followed up for 12 weeks after end of treatment.

Throughout the study, study visits will be conducted at the medical center and the patient's home. At certain planned study visits, patients will undergo a brief physical examination, and blood will be drawn for safety evaluation and for measuring biomarkers. At the Screening, Week 12, and Week 24 visits, patients will rate their disability and health-related quality of life using the Stroke Impact Scale. In addition, upper and lower extremity motor and sensory function (FMA-UE/LE), and gait velocity (Timed Up and Go) will be evaluated. Patients will be asked to report of any safety events throughout the study and follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-85 years
2. BMI: 18.0-35.0 kg/m2
3. Patient suffered an ischemic stroke (caused by blockage of the middle cerebral artery) 6-24 months prior to enrollment and with no additional symptomatic stroke incidents since then.
4. Patient resides in Israel between Hedera and Gedera
5. Fugl-Meyer Assessment of Upper Extremity: 20-50 without reflex items
6. Patient suffers from hemiparesis as assessed by the study investigator
7. Premorbid disability does not impact physical and cognitive function to a degree that would limit completion of study activities and assessments, as assessed by the study investigator
8. Patient agrees to participate in two physical therapy or occupational therapy sessions per week
9. Patient is able to use a device for telemedicine meetings with a physician and to record study-related events in an electronic diary, either alone or with caregiver's assistance

Exclusion Criteria:

1. Woman of childbearing potential who is pregnant or planning to become pregnant, or not using birth control
2. Aphasia or dementia limiting ability of patient to comply with instructions as assessed by the study investigator
3. Current diagnosis of severe depression (NOTE: In case of doubt, a patient who is currently taking or has taken within the last 30 days second-line anti-depressants OR who has scored 12-15 points using the Geriatric Depression Scale, will be considered severely depressed and will not be eligible to participate in the study.)
4. Drug or alcohol abuse within the last year
5. Current or planned Botox administration for upper limb spasticity, strabismus, overactive bladder, migraine prevention, blepharospasm, cervical dystonia or other off-label uses including but not limited to: sialorrhea, post-herpetic neuralgia, Raynaud's disease, achalasia, or any use the investigator believes may interfere with an accurate neurological exam. Permitted uses - cosmetic (wrinkles), hyperhidrosis
6. Participation in a transcranial magnetic stimulation and/or other interventional stroke studies within 6 months of screening
7. History of cancer within three years of screening, with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for at least 6 months
8. Any medical condition that, in the opinion of the investigator, would preclude patient participation in the study and/or analysis of results
9. Significant disability prior to stroke that would impact execution of any of the functional assessments in the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity (FM-UE) | 12 weeks
  Individual patient absolute change from baseline in motor and sensory functions as measured by the Fugl-Meyer Assessment of Upper Extremity (FMA-UE) 12 weeks after start of treatment.
Adverse Events | 12 weeks
  Incidence of adverse events (AEs) assessed according to CTCAE v5.0

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of Lower Extremity (FMA-LE) | 12 weeks
  Individual patient absolute change from baseline in motor and sensory functions as measured by the Fugl-Meyer Assessment of Lower Extremity (FMA-LE) 12 weeks after start of treatment.
Time Up and Go | 12 weeks
  Percent change from baseline gait velocity as measured by Timed Up and Go 12 weeks after start of treatment
Stroke Impact Scale | 12 weeks
  Absolute change from patient's baseline self-assessment as measured by Stroke Impact Scale 12 weeks after start of treatment, scored 0 to 100 with higher scores indicating higher quality of life
Durability of Fugl-Meyer | 24 weeks
  Absolute change in motor and sensory function as measured by the Fugl-Meyer Assessment of Upper and lower Extremity (FMA-UE & FMA-LE)
Durability of Time Up and Go | 24 weeks
  Percent change in gait velocity as measured by Timed Up and Go
Durability of Stroke Impact Scale | 24 weeks
  Absolute change in patient self-assessment as measured by Stroke Impact Scale over the 12-week follow-up period (12-24 weeks after the start of treatment); scored 0 to 100 with higher scores indicating higher quality of life

OTHER OUTCOMES:
Brain-derived neurotrophic factor (BDNF) | 12 weeks
  change in serum brain-derived neurotrophic factor
Neurofilament light chain (NfL) | 12 weeks
  change in serum neurofilament light chain

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No